CLINICAL TRIAL: NCT04716036
Title: Dissecting Responses to Alcohol in Individuals With Familial Risk for Bipolar Disorder
Brief Title: Familial Risk for Bipolar Disorder and Alcohol Sensitivity
Acronym: FACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Elizabeth Thomas Cox Lippard, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R21AA027884 (NIH)
Record Dates: First submitted 2021-01-12; First posted 2021-01-20 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Bipolar Disorder; Alcohol Drinking; Alcohol Use Disorder
MeSH Terms: conditions — Bipolar Disorder; Alcohol Drinking; Alcoholism | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol (Active Comparator): Participants will be dosed to a 0.08g% blood alcohol concentration.
  Interventions: Other: Alcohol beverage
- Placebo (Placebo Comparator): Participants will receive a low dose of alcohol (placebo condition).
  Interventions: Other: Placebo beverage

INTERVENTIONS:
Other: Alcohol beverage — Participants will be provided alcohol during study visits and changes in behavior/neural activity after consuming alcohol will be examined.
  Arms: Alcohol
Other: Placebo beverage — placebo beverage condition.
  Arms: Placebo

SUMMARY:
Early identification in individuals with bipolar disorder who are at risk for AUDs could inform novel intervention strategies and improve life-long outcomes. The primary objective of this protocol is to use alcohol administration procedures and alcohol biosensor technology to investigate responses to alcohol, compared to placebo, and relationship with parental risk for alcohol use disorders and/or bipolar disorder in young adults. Baseline clinical, cognitive, and behavioral assessments will be completed in 100 young adults (21-26 years; 50% women, no history of AUDs>mild). Participants would be equally divided among those with parental history of bipolar disorder but not AUDs, parental history of bipolar disorder and AUDs, parental history of AUDs but not bipolar disorder, and typically developing age- and sex-matched controls with no parental history of mood disorders or AUDs (N=25 per group). Then, while wearing Secure Continuous Remote Alcohol Monitoring [SCRAM] sensors, participants will complete within-person, counter-balanced, beverage sessions (following standard beverage administration procedures) in a simulated bar laboratory. Changes in heart rate, body sway and subjective self-report measurements of intoxication will also be completed while under the influence of alcohol or placebo. Specifically, individual differences in transdermal alcohol concentration (the primary data output from SCRAM sensors), physiological changes (e.g. heart rate), and the experience of stimulating, sedative, and anxiolytic effects of alcohol (measured with self-report surveys) will be investigated and differences between parental risk subgroups and healthy comparison participants investigated. Differences in transdermal alcohol concentration collected while under the influence of alcohol will be the primary data outcome assessed. Changes in heart rate, body sway, and experience of stimulating, sedative, and anxiolytic effects (from self-report survey data) while under the influence of alcohol compared to placebo session will also be investigated. Additionally, associations between objective and subjective responses to alcohol and drinking patterns will be explored (secondary outcome). The primary endpoint of the study will be after completion of both alcohol and placebo beverage conditions.

DETAILED DESCRIPTION:
A total of 100 young adults (21-26 years; 50% women, no history of AUDs>mild) will be recruited from the greater Austin area. Participants will be equally divided among those with parental history of bipolar disorder but not AUDs, parental history of bipolar disorder and AUDs, parental history of AUDs but not bipolar disorder, and typically developing age- and sex-matched controls with no parental history of mood disorders or AUDs (N=25 per group). The phone screen used for this study will assess parental history and clinical symptoms to achieve these recruitment goals for each subgroup.

Once recruited and enrolled, subjects will undergo detailed structured clinical evaluations to verify inclusion and exclusion criteria (including family history), comprehensive assessment of alcohol and other drug use history, and cognitive testing. Participants will return to the laboratory on subsequent days and complete their alcohol/placebo sessions while wearing Secure Continuous Remote Alcohol Monitoring (SCRAM) sensors and under the influence of alcohol or a placebo condition (counter-balanced). Following standard beverage administration procedures in a simulated bar laboratory, changes in heart rate, body sway, and self-report measures of subjective response to alcohol will be measured. Up to four participants will complete the beverage session together in the bar laboratory. This increases the ecological validity and strengthens the placebo manipulation. It also increases subject flow. Participants will be escorted to a private assessment room for all behavioral assessments. For each participant the first beverage session assignment (whether the participant is given alcohol or the placebo beverage first) will be randomized. The SCRAM sensor will be worn continuously and measure transdermal alcohol concentration throughout the alcohol and placebo sessions. Participants will wear the SCRAM sensor home overnight following their alcohol session and return the next morning for SCRAM sensor removal. Transdermal alcohol concentration is continuously collected overnight following an alcohol session. Participants will not be required to wear the SCRAM sensor home after their placebo session. For the placebo session, we will inform participants they received a low dose of alcohol and that their BrAC is at 0.0g% at the end of the session so monitoring overnight is not needed. Alcohol and placebo sessions will occur within 3 days of each other.

For both the alcohol and the placebo beverage conditions, the protocol will be the same. The beverage administration sessions will in a simulated bar laboratory in co-Investigator, Kim Fromme's, research suite at the University of Texas at Austin. The table in the testing room will be wiped down with alcohol prior to the participant's arrival (olfactory cue). Study staff will use an algorithm to calculate individual alcohol doses based on the participants' age, sex, height, and weight. Participants fast from food for 4 hours prior to their session. Before beginning consumption of their beverages, they will eat a weight-adjusted, 1 calorie per pound snack of pretzels. While participants eat their pretzels, study staff will mix beverages in front of participants. Vodka and placebo (decarbonated tonic water) will be stored in absolute vodka bottles, measured out, and combined with mixer in front of participants. Mixed drinks will be poured into glasses that have been sitting face down with rims soaking in vodka. Prior to giving the beverage to the participant, all drinks will get an alcohol floater (squirt of absolute vodka on top of the drink). Participants will be given 20 minutes to orally consume two beverages (10 minutes per beverage).

Following oral consumption and a 15-minute absorption period, breathalyzer tests will be conducted every 10 minutes to identify a .06g% ascending limb breath alcohol concentration (BrAC). Heart rate, body sway, and self-report of response to alcohol will be collected. BrAC will be measured at approximate 10 minute intervals, and heart rate, body sway, and subjective response to alcohol collected again at peak BrAC (0.08g%) and at descending BrAC of .06g%. Baseline heart rate, body sway, and self-report response (with instructions modified to ask how participants feel when they first arrive to the laboratory) are also collected before sessions begin so change on test days (e.g. peak 0.08g% BrAC heart rate - baseline heart rate) is calculated. Consistent with NIAAA guidelines for human alcohol studies, BrAC readings will continue every 30 minutes until participants are below 0.04% at which time they are escorted home. During the placebo condition, participants are told they will receive varying doses of alcohol, provided ambient olfactory cues, the rims of glasses are soaked in vodka, and alcohol floater is added to beverages (gustatory cues). A placebo manipulation test is measured during the ascending limb (placebo: after the absorption period with time of test given at the average time it takes individuals to reach ascending 0.06g% BrAC during the alcohol session) and when participants reach ascending 0.06g% BrAC (during alcohol session). Participants are asked to estimate the number of standard alcoholic drinks they were served. The average time participants stay in the laboratory will be shorter for the placebo vs. alcohol beverage condition. Participants are told they received a lower dose of alcohol and at the end of the placebo session they are told their BrAC is 0.0g%. They therefore do not need to wear the SCRAM sensor home. During the alcohol session participants are released at 0.04g% and they are told they need to wear the SCRAM sensor home overnight. Participants are debriefed, including BrAC reached during sessions, after they complete both sessions.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all participants:

* between 21 and 26 years of age
* having consumed at least 4 (men) or 3 (women) drinks on a single occasion at least twice over the last year
* euthymic at the time of study

Inclusion criteria for familial risk for bipolar disorder (only) participants:

- having at least one parent diagnosed with bipolar disorder type I, confirmed by family history interview

Inclusion criteria for familial risk for both bipolar disorder and alcohol use disorders participants:

* having at least one parent diagnosed with bipolar disorder type I, confirmed by family history interview
* having at least one parent diagnosed with an alcohol use disorder, confirmed by family history interview

Inclusion criteria for familial risk for alcohol use disorders (only) participants:

- having at least one parent diagnosed with an alcohol use disorder, confirmed by family history interview

Exclusion Criteria:

For all subjects exclusion criteria include:

* history of manic episode
* history of psychosis
* history of significant medical illness, particularly if possible changes in cerebral tissue
* full Scale IQ <85
* positive pregnancy test
* history of cannabis use disorder>moderate over past year
* history of AUD>mild over lifetime
* scores > 15 on the alcohol Use Disorders Identification Test (AUDIT; part of phone screen)
* ever being in an abstinence-oriented treatment program for alcohol use
* reporting wanting to quit drinking but not being able to
* any medical, religious, or other reasons for not drinking alcohol
* history of heart attack, heart trouble, high blood pressure, diabetes, or liver disease
* an adverse reaction to alcoholic beverages
* a flushing response (possibly suggesting altered alcohol metabolism)
* reporting never consuming 4 (men) or 3 (women) or more drinks on a single occasion at least twice over the last year
* unwillingness to have a friend or family member drive them home after the alcohol administration sessions
* a past substance use disorder (other than alcohol, cannabis, or nicotine) over the past year

Additional exclusion criteria for familial risk for bipolar disorder participants:

- not taking medications for >4 weeks (i.e. participants must be stable on antidepressant or anti-anxiety medication)

Additional exclusion criteria for healthy comparison subjects also include:

* any prior psychiatric hospitalizations
* lifetime history of a neurodevelopmental disorder, affective disorder, psychotic disorder, eating disorder
* having a parent diagnosed with a mood disorder or AUD
* greater than 1 month of lifetime psychotropic medication

Ages: 21 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in transdermal alcohol concentration: time to peak TAC | up to 24 hours
  Changes in transdermal alcohol concentration (TAC) during the alcohol session (i.e. time to reach peak TAC [measured in minutes]) will be compared between subgroups. Study participation to collect data (baseline clinical assessment, alcohol and placebo beverage sessions) should not take more than 13 hours. Participants will wear SCRAM sensors overnight following their alcohol session and return the following morning for SCRAM sensor removal (which takes <15 minutes).
Changes in transdermal alcohol concentration: peak TAC experienced | up to 24 hours
  Changes in transdermal alcohol concentration (TAC) during the alcohol session (i.e. peak TAC [g/dL]) will be compared between subgroups. Study participation to collect data (baseline clinical assessment, alcohol and placebo beverage sessions) should not take more than 13 hours. Participants will wear SCRAM sensors overnight following their alcohol session and return the following morning for SCRAM sensor removal (which takes <15 minutes).
Changes in transdermal alcohol concentration: area under the curve (AUC) | up to 24 hours
  Changes in transdermal alcohol concentration (TAC) during the alcohol session (i.e. geometric area under the curve [AUC]) will be compared between subgroups. Study participation to collect data (baseline clinical assessment, alcohol and placebo beverage sessions) should not take more than 13 hours. Participants will wear SCRAM sensors overnight following their alcohol session and return the following morning for SCRAM sensor removal (which takes <15 minutes).
  The units of the AUC are the units of the Y axis times units of the X axis. Y axis measures transdermal alcohol concentration in g/dL and the X axis measures time in minutes. The area is therefore expressed in units of (g/dL) x minutes.
Changes in transdermal alcohol concentration: absorption and elimination rates (g/dL per hour) | up to 24 hours
  Changes in transdermal alcohol concentration (TAC) during the alcohol session (i.e. absorption and elimination rates[g/dL per hour]) will be compared between subgroups. Study participation to collect data (baseline clinical assessment, alcohol and placebo beverage sessions) should not take more than 13 hours. Participants will wear SCRAM sensors overnight following their alcohol session and return the following morning for SCRAM sensor removal (which takes <15 minutes).
  Absorption rate is calculated as peak TAC (g/dL) divided by the time it took to rise from .000 to the peak; elimination rate is calculated as peak TAC divided by the time it took to decline from peak to .000 again.
Change (peak BrAC minus baseline BrAC) in heart rate will be compared between alcohol and placebo sessions. | up to 6 hours for alcohol session and up to 6 hours for placebo session
  Participants will have heart rate (beats per minute) measured they first arrive to both beverage administration sessions (alcohol and placebo). They will then have heart rate collected again during their beverage sessions (alcohol and placebo) at target BrACs (i.e, .08g%). Changes in heart rate will be calculated for both the alcohol and placebo conditions (i.e. at peak BrAC minus baseline BrAC) and compared.
Change (peak BrAC minus baseline BrAC) in body sway will be compared between alcohol and placebo sessions. | up to 6 hours for alcohol session and up to 6 hours for placebo session
  Participants will body sway measured when they first arrive to both beverage administration sessions (alcohol and placebo). They will then have body sway measured during their beverage sessions (alcohol and placebo) at target BrAC (.08g%). Changes in body sway will be calculated for both the alcohol and placebo conditions (i.e. at peak BrAC minus baseline BrAC) and compared.
Change (peak BrAC minus baseline BrAC) in behavior (self-report surveys) will be compared between alcohol and placebo sessions. | up to 6 hours for alcohol session and up to 6 hours for placebo session
  Participants will fill out self-report surveys (i.e., subjective effects of alcohol scale, drug effects questionnaire) on how they feel when they first arrive to both beverage administration sessions (alcohol and placebo). They will then fill out the same self-report surveys on how intoxicated they feel during their beverage sessions (alcohol and placebo) at target BrACs (i.e., .08g%). Changes in how intoxicated they feel will be calculated for both the alcohol and placebo conditions (i.e. at peak BrAC minus baseline BrAC) and compared.

SECONDARY OUTCOMES:
Recent alcohol use patterns relations with variability in transdermal alcohol concentration: time to reach peak TAC | baseline
  Participants will complete a structured assessment (time line follow back) to assess recent alcohol use including quantity (total drinks, average drinks per drinking day). Correlations between recent alcohol use and transdermal alcohol data (i.e. time to reach peak TAC [measured in minutes]) will be explored.
Recent alcohol use patterns relations with variability in transdermal alcohol concentration: peak TAC | baseline
  Participants will complete a structured assessment (time line follow back) to assess recent alcohol use including quantity (total drinks, average drinks per drinking day). Correlations between recent alcohol use and transdermal alcohol data (i.e. peak TAC [g/dL]) will be explored.
Recent alcohol use patterns relations with variability in transdermal alcohol concentration: area under the curve (AUC) | baseline
  Participants will complete a structured assessment (time line follow back) to assess recent alcohol use including quantity (total drinks, average drinks per drinking day). Correlations between recent alcohol use and transdermal alcohol data (i.e. geometric area under the curve [(g/dL) x minutes]) will be explored.
  The units of the AUC are the units of the Y axis times units of the X axis. Y axis measures transdermal alcohol concentration in g/dL and the X axis measures time in minutes. The area is therefore expressed in units of (g/dL) x minutes.
Recent alcohol use patterns relations with variability in transdermal alcohol concentration: absorption and elimination rates | baseline
  Participants will complete a structured assessment (time line follow back) to assess recent alcohol use including quantity (total drinks, average drinks per drinking day). Correlations between recent alcohol use and transdermal alcohol data (i.e. absorption and elimination rates [g/dL per hour]) will be explored.
  Absorption rate is calculated as peak TAC (g/dL) divided by the time it took to rise from .000 to the peak; elimination rate is calculated as peak TAC divided by the time it took to decline from peak to .000 again.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lippard, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
After study completion and publication of finding, transdermal alcohol concentration data and behavioral data collected following alcohol and placebo conditions will be shared.
Supporting Information: SAP
Time Frame: We will complete all our analyses and publish results and methodologies in scientific journals before the data are available to the research community. Data will be made available following 6 months after publication.
Access Criteria: We will be collecting identifying information. Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.